CLINICAL TRIAL: NCT01797445
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Versus Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Disoproxil Fumarate in HIV-1 Positive, Antiretroviral Treatment-Naïve Adults
Brief Title: Study to Evaluate the Safety and Efficacy of E/C/F/TAF Versus E/C/F/TDF in HIV-1 Positive, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-292-0111; 2013-000102-37 (EudraCT Number)
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2019-10

CONDITIONS: HIV; HIV Infections
Keywords: HIV; Treatment Naive; HIV 1 Infected; Women; Female
MeSH Terms: conditions — HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- E/C/F/TAF (Double-Blind) (Experimental): E/C/F/TAF plus E/C/F/TDF placebo for 144 weeks
  After 144 weeks, participants will continue to take their blinded study drug until treatment assignments have been unblinded.
  Interventions: Drug: E/C/F/TAF; Drug: E/C/F/TDF Placebo
- E/C/F/TDF (Double-Blind) (Active Comparator): E/C/F/TDF plus E/C/F/TAF placebo for 144 weeks
  After 144 weeks, participants will continue to take their blinded study drug until treatment assignments have been unblinded.
  Interventions: Drug: E/C/F/TDF; Drug: E/C/F/TAF Placebo
- Open-Label E/C/F/TAF (Experimental): After the unblinding visit, in countries where E/C/F/TAF is not commercially available, participants (except in UK) who complete 144 weeks of study will be given the option to receive open-label E/C/F/TAF and attend study visits every 12 weeks until it becomes commercially available, or until Gilead terminates the study in that country.
  Interventions: Drug: E/C/F/TAF

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablet administered orally once daily
  Other Names: Genvoya®
  Arms: E/C/F/TAF (Double-Blind); Open-Label E/C/F/TAF
Drug: E/C/F/TDF — 150/150/200/300 mg FDC tablet administered orally once daily
  Other Names: Stribild®
  Arms: E/C/F/TDF (Double-Blind)
Drug: E/C/F/TDF Placebo — Tablet administered orally once daily
  Arms: E/C/F/TAF (Double-Blind)
Drug: E/C/F/TAF Placebo — Tablet administered orally once daily
  Arms: E/C/F/TDF (Double-Blind)

SUMMARY:
The primary objective of this study is to evaluate the efficacy of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) fixed-dose combination (FDC) versus elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF) in HIV-1 positive, antiretroviral treatment-naive adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Plasma HIV-1 RNA levels ≥ 1,000 copies/mL at screening
* No prior use of any approved or investigational antiretroviral drug for any length of time, except the use for pre-exposure prophylaxis (PREP), or post-exposure prophylaxis (PEP) up to 6 months prior to screening
* Screening genotype report must show sensitivity to elvitegravir, emtricitabine, tenofovir DF
* Normal electrocardiogram (ECG)
* Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min according to the Cockcroft-Gault formula for creatinine clearance
* Hepatic transaminases (AST and ALT) ≤ 5 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Serum amylase ≤ 5 × ULN
* Males and females of childbearing potential must agree to utilize highly effective contraception methods or be non-heterosexually active or practice sexual abstinence from screening throughout the duration of study treatment and for 30 days following the last dose of study drug
* Females who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
* Females who have stopped menstruating for ≥ 12 months but do not have documentation of ovarian hormonal failure must have a serum follicle stimulating hormone (FSH) level at screening within the post-menopausal range based on the Central Laboratory reference range
* Age ≥ 18 years

Key Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to screening
* Hepatitis B surface antigen (HBsAg) positive
* Hepatitis C antibody positive
* Individuals experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance use judged by the Investigator to potentially interfere with study compliance
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements
* Participation in any other clinical trial (including observational trials) without prior approval
* Receiving ongoing therapy with drugs not to be used with elvitegravir, cobicistat, emtricitabine, tenofovir DF, and TAF or participants with any known allergies to the excipients of E/C/F/TDF or E/C/F/TAF

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 872 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2014-09-19 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (117):
- United States (79):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - Kaiser Permanente - Los Angeles Medical Center, Los Angeles, California
  - University of Southern California AIDS Clinical Trials Group, Los Angeles, California
  - Peter J. Ruane, Inc., Los Angeles, California
  - Anthony Mills MD Inc, Los Angeles, California
  - Alameda County Medical Center, Oakland, California
  - Stanford University, Palo Alto, California
  - University of California, Davis Medical Center, Sacramento, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Kaiser Permanente, San Leandro, California
  - Los Angeles Biomedical Research Institute at Harbor - UCLA Medical Center, Torrance, California
  - University of Colorado, Aurora, Colorado
  - APEX Research LLC, Denver, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Yale University, New Haven, Connecticut
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - Medical Faculty Associates, Washington D.C., District of Columbia
  - Gary J. Richmond,M.D.,P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - AIDS Healthcare Foundation, Miami, Florida
  - AIDS Healthcare Foundation, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Idocf/Valuhealthmd, Orlando, Florida
  - Infectious Diseases Associates of NW FL, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Infectious Disease Research Institute Inc., Tampa, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Atlanta ID Group, PC, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Infectious Disease Specialist of Atlanta, Decatur, Georgia
  - Mercer University, Macon, Georgia
  - University of Hawaii - Hawaii Center for AIDS, Honolulu, Hawaii
  - Rush University Medical Center, Section of Infectious Diseases, Chicago, Illinois
  - The Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Community Research Initiative of New England, Boston, Massachusetts
  - The Research Institute, West Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Central West Clinical Research, St Louis, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - ID Care, Hillsborough, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - Albany Medical College, Albany, New York
  - Upstate ID Assoc, Albany, New York
  - North Shore University Hospital - Division of Infectious Diseases, Manhasset, New York
  - Chelsea Village Medical, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina AIDS Clinical Trials Unit, Chapel Hill, North Carolina
  - Carolinas Medical Center Myer's Park Clinic, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University The Brody School of Medicine, Greenville, North Carolina
  - Rosedale Infectious Disseases, Huntersville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Central Texas Clinical Research, Austin, Texas
  - St. Hope Foundation, Inc., Bellaire, Texas
  - Trinity Health & Wellness Center / AIDS Arms, Inc., Dallas, Texas
  - Southwest Infectious Disease Clinical Research, Inc., Dallas, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon E. Crofoot, MD, PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education - Infectious Diseases (CARE-ID), Annandale, Virginia
  - Peter Shalit, MD, Seattle, Washington
- Canada (5):
  - Research Institute of McGill University Health Care, Montreal, Quebec
  - Clinique Medicale L'actuel, Montreal
  - University Health Network/Toronto General Hospital, Toronto
  - Maple Leaf Research, Toronto
  - Spectrum Health Care, Vancouver
- Instituto Dominicano de Estudios Virologicos--IDEV, Santo Domingo, Dominican Republic
- France (9):
  - Hopital de la Croix Rousse, Lyon
  - University Hospital of Montpellier (CHU-Gui de Chauliac), Montpellier
  - Archet 1 CHU de Nice, Department of Infectiology, Nice
  - Saint Louis Hospital of Infectious Diseases, Paris
  - Hopital Saint Antoine, Paris
  - Hôpital Bichat Claude Bernard, Paris
  - Hopital Tenon, Paris
  - Hopital Pitie Salpetriere, Paris
  - CH Tourcoing, Tourcoing
- Italy (2):
  - Universitaria di Bologna-Policlicnico S' Orsola Malpighi, Bologna
  - IRCCS Ospedale San Raffaele, Milan
- Mexico (2):
  - Hospital Civil de Guadalajara, Guadalajara
  - Insituto Nacional De Enfermedades Respiratorias "Ismael Cosio Villegas", Mexico City
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands
- Portugal (4):
  - Serviço de Doenças Infecciosas, HUC-CHUC, EPE, Coimbra
  - Hospital Santo Antonio dos Capuchos, Lisbon
  - Hospital de Santa Maria - CHLN, EPE, Lisbon
  - Centro Hospitalar do Porto - Hospital Joaquim Urbano, Porto
- Puerto Rico (2):
  - Hope Clinical Research, San Juan
  - University of Puerto Rico ACTU, San Juan
- Sweden (2):
  - Venhalsan / Sodersjukhuset, Stockholm
  - Karolinska University Hospital, Huddinge, Stockholm
- United Kingdom (10):
  - Whittall Street Clinic, Birmingham
  - Heart Of England NHS Foundation Trust, Birmingham
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Brownlee Centre, Gartnavel General Hospital, Glasgow
  - Barts Health NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Kings College Hospital, London
  - Chelsea and Westminster, London
  - Mortimer Market Centre, London
  - North Manchester General Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Sax PE, Wohl D, Yin MT, Post F, DeJesus E, Saag M, Pozniak A, Thompson M, Podzamczer D, Molina JM, Oka S, Koenig E, Trottier B, Andrade-Villanueva J, Crofoot G, Custodio JM, Plummer A, Zhong L, Cao H, Martin H, Callebaut C, Cheng AK, Fordyce MW, McCallister S; GS-US-292-0104/0111 Study Team. Tenofovir alafenamide versus tenofovir disoproxil fumarate, coformulated with elvitegravir, cobicistat, and emtricitabine, for initial treatment of HIV-1 infection: two randomised, double-blind, phase 3, non-inferiority trials. Lancet. 2015 Jun 27;385(9987):2606-15. doi: 10.1016/S0140-6736(15)60616-X. Epub 2015 Apr 15. PMID 25890673
- [Result] Margot N, Cox S, Das M, McCallister S, Miller MD, Callebaut C. Rare emergence of drug resistance in HIV-1 treatment-naive patients receiving elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide for 144 weeks. J Clin Virol. 2018 Jun;103:37-42. doi: 10.1016/j.jcv.2018.03.012. Epub 2018 Apr 2. PMID 29627709
- [Result] Arribas JR, Thompson M, Sax PE, Haas B, McDonald C, Wohl DA, DeJesus E, Clarke AE, Guo S, Wang H, Callebaut C, Plummer A, Cheng A, Das M, McCallister S. Brief Report: Randomized, Double-Blind Comparison of Tenofovir Alafenamide (TAF) vs Tenofovir Disoproxil Fumarate (TDF), Each Coformulated With Elvitegravir, Cobicistat, and Emtricitabine (E/C/F) for Initial HIV-1 Treatment: Week 144 Results. J Acquir Immune Defic Syndr. 2017 Jun 1;75(2):211-218. doi: 10.1097/QAI.0000000000001350. PMID 28282300
- [Result] Margot N, Cox S, Das M, McCallister S, Miller MD, Callebaut C. Infrequent development of drug resistance in HIV-1-infected treatment-naive subjects after 96 weeks of treatment with elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate. Antivir Ther. 2017;22(5):443-446. doi: 10.3851/IMP3125. Epub 2017 Jan 11. PMID 28076335
- [Result] Margot NA, Kitrinos KM, Fordyce M, McCallister S, Miller MD, Callebaut C. Rare emergence of drug resistance in HIV-1 treatment-naive patients after 48 weeks of treatment with elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide. HIV Clin Trials. 2016 Mar;17(2):78-87. doi: 10.1080/15284336.2016.1142731. PMID 26892863
- [Result] Funderburg NT, McComsey GA, Kulkarni M, Bannerman T, Mantini J, Thornton B, Liu HC, Zhang Y, Song Q, Fang L, Dinoso J, Cheng A, McCallister S, Fordyce MW, Das M. Equivalent Decline in Inflammation Markers with Tenofovir Disoproxil Fumarate vs. Tenofovir Alafenamide. EBioMedicine. 2016 Nov;13:321-327. doi: 10.1016/j.ebiom.2016.10.009. Epub 2016 Oct 11. PMID 27742226
- [Result] Wohl D, Oka S, Clumeck N, Clarke A, Brinson C, Stephens J, Tashima K, Arribas JR, Rashbaum B, Cheret A, Brunetta J, Mussini C, Tebas P, Sax PE, Cheng A, Zhong L, Callebaut C, Das M, Fordyce M; GS-US-2,92-01040111 and Study Team. Brief Report: A Randomized, Double-Blind Comparison of Tenofovir Alafenamide Versus Tenofovir Disoproxil Fumarate, Each Coformulated With Elvitegravir, Cobicistat, and Emtricitabine for Initial HIV-1 Treatment: Week 96 Results. J Acquir Immune Defic Syndr. 2016 May 1;72(1):58-64. doi: 10.1097/QAI.0000000000000940. PMID 26829661
- [Result] Custodio JM, Garner W, Callebaut C, Fordyce M, Plummer A, Zhong L, et al. The Pharmacokinetics of Tenofovir and Tenofovir Diphosphate Following Administration of Tenofovir Alafenamide vs Tenofovir Disoproxil Fumarate [Oral Abstract #6]. The 16th International Workshop on Clinical Pharmacology of HIV & Hepatitis Therapy. Washington DC, USA, May 26-28, 2015.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America and Europe. The first participant was screened on 12 March 2013. The last study visit occurred on 03 October 2018.
Pre-assignment Details: 1070 participants were screened.
Groups:
- E/C/F/TAF: Double-Blind Phase: Elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablet plus elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF) placebo tablet administered orally once daily for 144 weeks.
  Open-Label Extension Phase: After the unblinding visit, in countries where E/C/F/TAF FDC was not commercially available, participants (except in UK) were given the option to receive the open-label E/C/F/TAF FDC until it became commercially available, or until Gilead terminated the study in that country.
- E/C/F/TDF: Double-Blind Phase: E/C/F/TDF (150/150/200/300 mg) FDC tablet plus E/C/F/TAF placebo tablet administered orally once daily for 144 weeks.
  Open-Label Extension Phase: After the unblinding visit, in countries where E/C/F/TAF FDC was not commercially available, participants (except in UK) were given the option to receive the open-label E/C/F/TAF FDC until it became commercially available, or until Gilead terminated the study in that country.
Period: Double-Blind Phase
Arm/Group | E/C/F/TAF | E/C/F/TDF
Started | 435 | 437
Completed | 348 | 348
Not Completed | 87 | 89
Not completed — Randomized but Not Treated | 4 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Death | 5 | 4
Not completed — Pregnancy | 0 | 1
Not completed — Lack of Efficacy | 1 | 2
Not completed — Investigator's Discretion | 15 | 17
Not completed — Noncompliance with Study Drug | 5 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrew Consent | 20 | 35
Not completed — Lost to Follow-up | 34 | 26
Period: Open-Label Extension Phase
Arm/Group | E/C/F/TAF | E/C/F/TDF
Started | 141 (207 participants completed the Double-Blind Phase, but did not enter the Open-Label Extension Phase.) | 119 (229 participants completed the Double-Blind Phase, but did not enter the Open-Label Extension Phase.)
Completed | 140 | 119
Not Completed | 1 | 0
Not completed — Investigator's Discretion | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- E/C/F/TAF: E/C/F/TAF (150/150/200/10 mg) FDC tablet plus E/C/F/TDF placebo tablet administered orally once daily for 144 weeks
- E/C/F/TDF: E/C/F/TDF (150/150/200/300 mg) FDC tablet plus E/C/F/TAF placebo tablet administered orally once daily for 144 weeks
- Total: Total of all reporting groups
Arm/Group | E/C/F/TAF | E/C/F/TDF | Total
Number analyzed (Participants) | 431 | 435 | 866
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10.8) | 36 (10.9) | 36 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 71 | 133
  Male | 369 | 364 | 733
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 15 | 12 | 27
  Black | 129 | 132 | 261
  Native Hawaiian or Pacific Islander | 4 | 1 | 5
  White | 235 | 243 | 478
  Other | 47 | 44 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 107 | 97 | 204
  Not Hispanic or Latino | 323 | 336 | 659
  Not Permitted | 1 | 1 | 2
  Missing | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 280 | 282 | 562
  United Kingdom | 25 | 31 | 56
  Portugal | 21 | 16 | 37
  Canada | 19 | 22 | 41
  Netherlands | 6 | 8 | 14
  Sweden | 8 | 3 | 11
  Dominican Republic | 30 | 35 | 65
  Italy | 10 | 8 | 18
  Mexico | 16 | 12 | 28
  France | 16 | 18 | 34
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.53 (0.647) | 4.50 (0.690) | 4.52 (0.669)
HIV-1 RNA Category [Count of Participants; unit: Participants]
  ≤ 100,000 copies/mL | 339 | 336 | 675
  > 100,000 to ≤ 400,000 copies/mL | 68 | 82 | 150
  > 400,000 copies/mL | 24 | 17 | 41
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] — Population: Participants in the Safety Analysis Set with available data were analyzed (E/C/F/TAF: N = 430; E/C/F/TDF: N = 435)
  cells/µL
    number analyzed (Participants) | 430 | 435 | 865
    (all) | 414 (206.8) | 431 (226.8) | 423 (217.1)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  < 50 cells/μL | 14 | 15 | 29
  ≥ 50 to < 200 cells/μL | 40 | 49 | 89
  ≥ 200 to < 350 cells/μL | 115 | 89 | 204
  ≥ 350 to < 500 cells/μL | 134 | 149 | 283
  ≥ 500 cells/μL | 127 | 133 | 260
  Missing | 1 | 0 | 1
HIV Disease Status [Count of Participants; unit: Participants]
  Asymptomatic | 377 | 394 | 771
  Symptomatic HIV Infection | 30 | 19 | 49
  AIDS | 22 | 19 | 41
  Unknown | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: The Full Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 431 | 435
percentage of participants | 91.6 | 88.5
Statistical Analysis 1: Comparison: E/C/F/TAF vs E/C/F/TDF; Null hypothesis: the E/C/F/TAF group was ≥ 12% worse than the E/C/F/TDF group with respect to the percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48; alternative hypothesis: the E/C/F/TAF group was < 12% worse than the E/C/F/TDF group; Test type: Superiority or Other; p = 0.13, Cochran-Mantel-Haenszel; P-value was from the Cochran-Mantel-Haenszel (CMH) test stratified by baseline HIV-1 RNA (≤ 100,000 or > 100,000 copies/mL) and region (US vs ex-US); Difference in Percentages = 3.1, 95.002% CI 2-sided [-1.0 to 7.1] — The difference in percentages and its 95.002% confidence interval (CI) were calculated based on the Mantel-Haenszel (MH) proportions adjusted by baseline HIV-1 RNA and region stratum

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 431 | 435
percentage of participants | 84.0 | 82.3

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Weeks 48 and 96
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Weeks 48 and 96 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Weeks 48 and 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 431 | 435
percentage of participants
  Week 48 | 82.4 | 80.7
  Week 96 | 78.7 | 76.8

4. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 404 | 400
cells/µL | 225 (171.2) | 200 (162.5)

5. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 369 | 369
cells/µL | 274 (184.0) | 260 (179.6)

6. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Description: Hip BMD was assessed by dual energy x-ray absorptiometry (DXA) scan.
Time Frame: Baseline; Week 48
Population: The Hip DXA Analysis Set included all participants who were randomized and received at least 1 dose of study drug, and have nonmissing baseline hip BMD values. Participants were grouped according to the treatment they actually received. The missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 380 | 381
percent change | -0.420 (3.2268) | -2.603 (3.1482)

7. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 96
Description: Hip BMD was assessed by DXA scan.
Time Frame: Baseline; Week 96
Population: Participants in the Hip DXA Analysis Set were analyzed. Participants were grouped according to the treatment they actually received. The missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 341 | 346
percent change | -0.364 (3.8990) | -3.023 (3.9796)

8. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 48
Population: The Spine DXA Analysis Set included all participants who were randomized and received at least 1 dose of study drug, and have nonmissing baseline spine BMD values. Participants were grouped according to the treatment they actually received. The missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 386 | 385
percent change | -1.278 (3.0098) | -2.759 (3.0024)

9. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 96
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 96
Population: Participants in the Spine DXA Analysis Set were analyzed. Participants were grouped according to the treatment they actually received. The missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 346 | 347
percent change | -1.017 (3.3957) | -2.516 (3.8612)

10. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 48
Time Frame: Baseline; Week 48
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug. The missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 405 | 402
mg/dL | 0.08 (0.136) | 0.12 (0.283)

11. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set were analyzed. The missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 373 | 370
mg/dL | 0.04 (0.119) | 0.07 (0.122)

12. Secondary Outcome: Percentage of Participants With Treatment-emergent Proteinuria Through Week 48
Description: Grades 1 (mild), 2 (moderate), and 3 (severe) were the highest treatment-emergent postbaseline grades for urine protein using the dipstick method. The worst postbaseline value is presented for each participant.
Time Frame: Baseline to Week 48
Population: Participants in the Safety Analysis Set with at least 1 postbaseline urine protein value were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 428 | 434
percentage of participants
  Grade 1 | 27.3 | 31.6
  Grade 2 | 4.7 | 4.6
  Grade 3 | 0 | 0

13. Secondary Outcome: Percentage of Participants With Treatment-emergent Proteinuria Through Week 96
Description: as for outcome 12
Time Frame: Baseline to Week 96
Population: Participants in the Safety Analysis Set with at least 1 postbaseline urine protein value were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 428 | 434
percentage of participants
  Grade 1 | 31.8 | 36.9
  Grade 2 | 5.4 | 5.1
  Grade 3 | 0 | 0

14. Secondary Outcome: Percent Change From Baseline in Urine Retinol Binding Protein (RBP) to Creatinine Ratio at Week 48
Description: Urine RBP is a renal biomarker which is used to detect drug-induced kidney injury.
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 400 | 397
percent change | 13.3 [-22.6 to 52.4] | 51.7 [2.6 to 138.6]

15. Secondary Outcome: Percent Change From Baseline in Urine RBP to Creatinine Ratio at Week 96
Description: Urine RBP is a renal biomarker which is used to detect drug-induced kidney injury.
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 379 | 363
percent change | 16.9 [-18.6 to 72.4] | 73.7 [10.4 to 196.3]

16. Secondary Outcome: Percent Change From Baseline in Urine Beta-2-microglobulin to Creatinine Ratio at Week 48
Description: Urine Beta-2-microglobulin is a renal biomarker which is used to detect drug-induced kidney injury.
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 395 | 392
percent change | -29.3 [-55.1 to 6.1] | 32.3 [-36.4 to 159.9]

17. Secondary Outcome: Percent Change From Baseline in Urine Beta-2-microglobulin to Creatinine Ratio at Week 96
Description: Urine Beta-2-microglobulin is a renal biomarker which is used to detect drug-induced kidney injury.
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | E/C/F/TAF | E/C/F/TDF
Number analyzed (Participants) | 375 | 360
percent change | -31.0 [-62.7 to 6.1] | 35.2 [-27.5 to 248.8]

ADVERSE EVENTS:
Time Frame: First dose date to last dose date (maximum duration: 185 weeks during Double-Blind Phase and 102 weeks during Open-Label Extension Phase) plus 30 days
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- E/C/F/TAF (Double-Blind Phase): Adverse events reported occurred during the Double-Blind Phase in participants from the E/C/F/TAF group, who received E/C/F/TAF (150/150/200/10 mg) FDC tablet plus E/C/F/TDF placebo tablet administered orally once daily for 144 weeks.
- E/C/F/TDF (Double-Blind Phase): Adverse events reported occurred during the Double-Blind Phase in participants from the E/C/F/TDF group, who received E/C/F/TDF (150/150/200/300 mg) FDC tablet plus E/C/F/TAF placebo tablet administered orally once daily for 144 weeks.
- Open-Label E/C/F/TAF From E/C/F/TAF: Adverse events reported occurred during the Open-Label Extension Phase in participants who enrolled into the Open-Label Extension Phase from the E/C/F/TAF group and received E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily.
- Open-Label E/C/F/TAF From E/C/F/TDF: Adverse events reported occurred during the Open-Label Extension Phase in participants who enrolled into the Open-Label Extension Phase from the E/C/F/TDF group and received E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily.
Arm/Group | E/C/F/TAF (Double-Blind Phase) | E/C/F/TDF (Double-Blind Phase) | Open-Label E/C/F/TAF From E/C/F/TAF | Open-Label E/C/F/TAF From E/C/F/TDF
All-Cause Mortality (participants affected / at risk) | 5/431 | 4/435 | 0/141 | 0/119
Serious Adverse Events (participants affected / at risk) | 54/431 | 68/435 | 4/141 | 2/119
Other Adverse Events (participants affected / at risk) | 374/431 | 366/435 | 32/141 | 27/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (Double-Blind Phase) (N=431) | E/C/F/TDF (Double-Blind Phase) (N=435) | Open-Label E/C/F/TAF From E/C/F/TAF (N=141) | Open-Label E/C/F/TAF From E/C/F/TDF (N=119)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Palatal dysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 3 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 2 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 2 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 4 | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 0 | 0
Chorioretinitis (Infections and infestations) | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0
Infectious colitis (Infections and infestations) | 0 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis meningococcal (Infections and infestations) | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Penile abscess (Infections and infestations) | 1 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 2 | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Scrotal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Secondary syphilis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Shigella infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 2 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 1 | 0 | 0
West Nile viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Labelled drug-drug interaction medication error (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase abnormal (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Bipolar II disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 3 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 2 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 2 | 0 | 0
Renal haematoma (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 0
Vaginal dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (Double-Blind Phase) (N=431) | E/C/F/TDF (Double-Blind Phase) (N=435) | Open-Label E/C/F/TAF From E/C/F/TAF (N=141) | Open-Label E/C/F/TAF From E/C/F/TDF (N=119)
Lymphadenopathy (Blood and lymphatic system disorders) | 29 | 24 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 33 | 34 | 0 | 2
Constipation (Gastrointestinal disorders) | 24 | 33 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 99 | 114 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 23 | 15 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 26 | 27 | 1 | 1
Nausea (Gastrointestinal disorders) | 78 | 86 | 1 | 2
Toothache (Gastrointestinal disorders) | 26 | 19 | 1 | 1
Vomiting (Gastrointestinal disorders) | 44 | 46 | 0 | 2
Fatigue (General disorders) | 53 | 52 | 1 | 0
Pyrexia (General disorders) | 37 | 32 | 0 | 0
Bronchitis (Infections and infestations) | 38 | 26 | 2 | 1
Chlamydial infection (Infections and infestations) | 24 | 20 | 1 | 0
Folliculitis (Infections and infestations) | 19 | 26 | 2 | 0
Gastroenteritis (Infections and infestations) | 23 | 21 | 0 | 2
Gonorrhoea (Infections and infestations) | 26 | 20 | 1 | 0
Influenza (Infections and infestations) | 25 | 18 | 1 | 2
Nasopharyngitis (Infections and infestations) | 68 | 75 | 5 | 5
Pharyngitis (Infections and infestations) | 22 | 25 | 0 | 0
Sinusitis (Infections and infestations) | 25 | 28 | 2 | 1
Syphilis (Infections and infestations) | 42 | 44 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 87 | 82 | 2 | 2
Urinary tract infection (Infections and infestations) | 17 | 31 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 61 | 49 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 63 | 53 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 34 | 38 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 | 26 | 2 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 29 | 25 | 0 | 1
Dizziness (Nervous system disorders) | 27 | 28 | 1 | 0
Headache (Nervous system disorders) | 98 | 80 | 4 | 2
Anxiety (Psychiatric disorders) | 34 | 43 | 0 | 0
Depression (Psychiatric disorders) | 34 | 26 | 0 | 1
Insomnia (Psychiatric disorders) | 51 | 37 | 1 | 0
Proteinuria (Renal and urinary disorders) | 11 | 22 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 62 | 49 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16 | 22 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 39 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 47 | 42 | 1 | 0
Hypertension (Vascular disorders) | 26 | 11 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years